CLINICAL TRIAL: NCT01189331
Title: Non-invasive Functional Assessment of Coronary Stenoses Using CT Coronary Angiography and Computational Fluid Dynamics
Brief Title: CT Coronary Angiography and Computational Fluid Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University (Other); Pauls Stradins Clinical University Hospital (Other); Cornell University (Other); Ulsan university (Unknown); Indiana University (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1007-193-325
Record Dates: First submitted 2010-08-15; First posted 2010-08-26 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; CT; Computational flow dynamics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: With masking value of FFR derived from coronary CT angiography to the investigators, FFR is measured and patients have been followed-up.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT and FFR (No Intervention)
  Interventions: Device: CT coronary angiography and computational fluid dynamics

INTERVENTIONS:
Device: CT coronary angiography and computational fluid dynamics — Evaluate coronary blood flow dynamics by CT coronary angiography and computational fluid dynamics

SUMMARY:
Angiographically obtained fractional flow reserve(FFR) could provide functional and clinical information about stenotic lesion, but the invasiveness and measuring difficulty of FFR make it unfamiliar to perform. CT coronary angiography is non-invasive tool to evaluate lesion severity and lately developing computational fluid dynamics could provide functional information. The investigators build a patient specific model of computational fluid dynamics by CT coronary angiography and evaluate the functional significance by measuring fractional flow reserve via CT coronary angiography and computational fluid dynamics, and investigate its long-term prognostic implications.

ELIGIBILITY:
Inclusion Criteria:

* Significant stenosis at CT angiography
* Normal ejection fraction on echocardiography
* Informed consented patient

Exclusion Criteria:

* total occlusion and collateral flow to target vessel
* AV conduction abnormality
* Left ventricular hypertrophy
* significant valvular heart or primary myocardial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-10-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
fractional flow reserve | 1day
  fractional flow reserve of stenotic coronary artery
target vessel failure | 10 year
  composite of cardiovascular death, target vessel myocardial infarction, target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yang S, Chung J, Lesina K, Doh JH, Jegere S, Erglis A, Leipsic JA, Fearon WF, Narula J, Koo BK. Long-term prognostic implications of CT angiography-derived fractional flow reserve: Results from the DISCOVER-FLOW study. J Cardiovasc Comput Tomogr. 2024 May-Jun;18(3):251-258. doi: 10.1016/j.jcct.2024.01.016. Epub 2024 Feb 19. PMID 38378313
- [Derived] Yang S, Lesina K, Doh JH, Jegere S, Erglis A, Leipsic JA, Chun EJ, Choi G, Schaap M, Zarins C, Taylor CA, Fearon WF, Narula J, Koo BK. Long-term prognostic implications of hemodynamic and plaque assessment using coronary CT angiography. Atherosclerosis. 2023 May;373:58-65. doi: 10.1016/j.atherosclerosis.2023.02.005. Epub 2023 Feb 27. PMID 36872186
- [Derived] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711